CLINICAL TRIAL: NCT02360514
Title: Non-comparable and Open Clinical Research to Evaluate Long-term Immunity by Neutralizing Antibody Test of Adults in High Risk Population of HFRS (Hemorrhagic Fever With Renal Syndrome) After Vaccination and Booster Vaccination of Hantavax
Brief Title: Study to Evalutate Long-term Immunity of Hantavax in High Risk Population of HFRS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HTV_P3
Record Dates: First submitted 2015-02-03; First posted 2015-02-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- hantaan virus vaccine (Experimental)
  Interventions: Drug: Hantavax injection

INTERVENTIONS:
Drug: Hantavax injection — Intramuscular or hypodermic injection of 0.5ml per time twice at interval of 1 month for adults. For more immune, inoculate muscle or subcutaneous once mor 12 months after the completion of the initial immune

SUMMARY:
This study was aimed evaluate long-term immunity response by neutralizing antibody test of adults in high risk population of HFRS .

DETAILED DESCRIPTION:
This clinical trial was designed as a multicenter, non-comparable, open-label clinical trial.This trial was conducted written informed consent form by voluntary agreement, negative result of hantaanvirus antubidy by neutralizaing antibody test, test drug was administrated 0, 1, 13 months according to drug label.

For antibody test, Sampling was conducted pre-dose(T0), 1 month after vaccination(T1), 1 year after vaccination(before booster vaccination, T2) and 1 month after vaccination(T3). Also, 1 month after vaccination (T3) after completion of booster vaccination for antibody retension duration observed for subjects with antibody to conduct a three-year follow-up survey was conducted, and the antibody test every year.In conclusion, sampling was conducted 12 months(T4), 24 months(T5), 36months(T6) after the booster vaccionation.

However, follow-up survey was terminated when the antibody titer was determined as a negative by neutralizing antibody test and fluorescent antibody technique.

ELIGIBILITY:
Inclusion Criteria:

* The subjects who have the vaccination history of ah the time of screening
* The subjects whose Hantaan virus virus's antibody shows negative using Neutralizing antibody test at the time of screening

Exclusion Criteria:

* The subjects who have a history of hemorrhagic fever with renal syndrome
* The subjects who have a fever or significant dystrophy

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2007-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Antibody seroconversion rates at 1 month after the booster vaccination and its retention rates | 13 months

SECONDARY OUTCOMES:
The antibody seroconversion rates and its retension rates by neutralizing antibody test | 13 months
  After vaccination (2 times) and booster vaccination (1 time) of Hantavax to adults in high risk population
The antibody seroconversion rates and its retension rates by fluorescent antibody technique | 13 months
  After vaccination (2 times) and booster vaccination (1 time) of Hantavax to adults in high risk population
The antibody titers by neutralizing antibody test and fluorescent antibody technique | 13 months
Number of adverse events after vaccination of Hantavax to adults in high risk population. | 3 years